CLINICAL TRIAL: NCT02336256
Title: Plasma Total Antioxidant Status and Thiobarbituric Acid-reacting Substances in Patients With Inguinal Hernia Operated by Totally Extraperitoneal (TEP) or Single Incision Laparoscopic Surgery (SILS)
Brief Title: Plasma Total Antioxidant Status and Thiobarbituric Acid-reacting Substances in Patients With Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jacek Białecki, MD, PhD, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JB-1
Record Dates: First submitted 2014-12-16; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia repair; totally extraperitoneal (TEP); single incision laparoscopic surgery (SILS); plasma total antioxidant status
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEP SILS (Experimental): Procedures of hernia repair. Patients operated due to inguinal hernia using modified single incision laparoscopic surgery (SILS) methods.
  Interventions: Procedure: Procedures of hernia repair.
- Typical TEP (Active Comparator): Procedures of hernia repair. Patients operated due to inguinal hernia using typical totally extra peritoneal.
  Interventions: Procedure: Procedures of hernia repair.

INTERVENTIONS:
Procedure: Procedures of hernia repair. — We use two procedure: single incision laparoscopic surgery (SILS) and totally extra-peritoneal repair (TEP). SILS procedure used one approche - 10mm (experimental). TEP procedure used three approaches 2x5mm and 1x10mm (active comparator).

SUMMARY:
Introduction: Any form of trauma, including surgery is known to result in oxidative stress. Single incision laparoscopy is a step forward towards almost scarless surgery. It is also expected to result in a lower degree of free radicals generation and faster normalization of the organism's antioxidant capacity.

Aim: The aim of the study was to assess a number of plasma oxidative stress markers in patients operated due to inguinal hernia using typical totally extra peritoneal (TEP) and modified single incision laparoscopic surgery (SILS) methods.

Material and methods: Thirty-two consecutive patients with no acute disease and severe chronic disorder, were qualified for inguinal hernia laparoscopic surgery. All were caucasian males, aged 24-69 and they underwent one of two surgical approaches: totally extra-peritoneal repair (TEP) and single incision laparoscopic surgery (SILS). TEP patients created Group 1 (n= 17) and SILS patients formed Group 2 (n= 17). Total antioxidant status (TAS) and thiobarbituric acid-reacting substances (TBARS) were determined in three time points: before, one day and four days after the laparoscopic surgery.

DETAILED DESCRIPTION:
Thirty-two consecutive patients with no acute disease and severe chronic disorder were qualified for inguinal hernia laparoscopic surgery. All were caucasian males, aged 24-69 underwent one of two different surgical approaches: totally extra-peritoneal (TEP) repair and single incision laparoscopic surgery (SILS). TEP patients created Group 1 (n= 17) and SILS patients formed Group 2 (n= 17).

Blood Sampling and Biochemical Analysis Ulnar venous blood samples were collected from the participants three times (fasting, between 6:00 and 7:00 AM): before (0), one day (1) and four days (2) after laparoscopic surgery. Baseline (0) blood samples were used for routine pre-operative laboratory assessment, including complete blood count, basic coagulation tests, C-reactive protein, glucose and electrolytes levels. Total antioxidant status (TAS) and thiobarbituric acid-reacting substances (TBARS) were determined in three time points: 0, 1 and 2 as described above.

Spectrophotometry was used to measure TAS (RANDOX Laboratories, Crumlin, Antrim, UK) on Statfax 1904Plus (Awareness Technology, Palm City, FL) and TBARS according to the Okhawa method [11] (Sigma reagents, Germany) on Specord M40 (Carl-Zeiss, Germany). The intra- and inter-assay coefficients of variation were as follows: TAS (1.6 % and 3.7%), and TBARS (1.9% and 3.8%)

ELIGIBILITY:
Inclusion Criteria:

* Patients with inguinal hernia.

Exclusion Criteria:

* Patients with acute disease and severe chronic disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the concentration of Total antioxidant status, Thiobarbituric acid-reacting substances. | Before treatment

SECONDARY OUTCOMES:
Assessment of changes in the concentration of Total antioxidant status, Thiobarbituric acid-reacting substances. | One day after the laparoscopic surgery

OTHER OUTCOMES:
Assessment of changes in the concentration of Total antioxidant status, Thiobarbituric acid-reacting substances. | Four days after the laparoscopic surgery